CLINICAL TRIAL: NCT00362531
Title: Phase 3 Study of Tacrolimus Combined With Prednisone Treatment of Idiopathic Membranous Nephropathy and Nephrotic Syndrome
Brief Title: Tacrolimus Combined With Prednisone Treatment of Idiopathic Membranous Nephropathy and Nephrotic Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Peking University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRGNSCN01-0; NCT00268567
Record Dates: First submitted 2006-08-09; First posted 2006-08-10 (Estimated); Last update posted 2006-08-10 (Estimated); Status verified 2006-01

CONDITIONS: Idiopathic Membranous Nephropathy; Nephrotic Syndrome
MeSH Terms: conditions — Glomerulonephritis, Membranous; Nephrotic Syndrome | interventions — Prednisone

INTERVENTIONS:
Drug: tacrolimus combined with prednisone

SUMMARY:
Idiopathic membranous nephropathy (IMN) is one of the most common forms of nephrotic syndrome (NS) in adults and is usually treated by corticosteroids in combination with cytotoxic drugs especially cyclophosphamide or cyclosporine. Tacrolimus, a new immunosuppressive agent, was proved to be effective in treating refractory NS. Whether it is effective in IMN has not been reported. We therefore undertook a multi-center, controlled study to investigate the efficacy and safety profile of tacrolimus compared with cyclophosphamide in the treatment of patients with idiopathic membranous nephropathy and nephrotic syndrome.

DETAILED DESCRIPTION:
Idiopathic membranous nephropathy (IMN) is one of the most common forms of nephrotic syndrome (NS) in adults and is usually treated by corticosteroids in combination with cytotoxic drugs especially cyclophosphamide or cyclosporine. However, the effect was not satisfying and the side-effects of the above immunosuppressive agents were often a worrying problem. Tacrolimus, a new immunosuppressive agent, was proved to be effective in treating refractory NS especially FSGS. Whether it is effective in IMN has not been reported. We therefore undertook a multi-center, controlled study to investigate the efficacy and safety profile of tacrolimus compared with cyclophosphamide in the treatment of patients with idiopathic membranous nephropathy and nephrotic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* All patients were diagnosed as idiopathic membranous nephropathy according to renal histology, with nephrotic syndrome, serum creatinine less than 2.5mg/dL, 18~70 years old, signed the informed consent and willing to be followed up according to the protocol.

Exclusion Criteria:

* Patients who had received immunosuppressive therapy within the previous 3 months, complicated other severe renal diseases, serum creatinine higher than 2.5mg/dL, severe infection, diabetes mellitus, liver disease, pregnancy, lactating, and anticipated poor compliance with the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-11; Study Completion 2007-01

PRIMARY OUTCOMES:
complete remission of renal disease at 12 months

SECONDARY OUTCOMES:
partial remission at 12 months and adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan WANG, MD, Principal Investigator — Renal Division, Peking University First Hospital; Jianghua Chen, MD, Principal Investigator — Department of Nephrology, First Hospital of Zhejiang University; Xuewang Li, MD, Principal Investigator — Department of Nephrology, Peking Union Medical College Hospital; Fuming Lu, MD, Principal Investigator — Department of Nephrology, Huashan Hospital, Fudan University; Feifei Xu, MD, Principal Investigator — Department of Nephrology, First Hospital of Wenzhou Medical College; Jiaqi Qian, MD, Principal Investigator — Department of Nephrology, Renji Hospital of Shanghai; Fanfan Hou, MD, Principal Investigator — Department of Nephrology, Nanfang Hospital, First Military Medical University

REFERENCES:
- [Derived] von Groote TC, Williams G, Au EH, Chen Y, Mathew AT, Hodson EM, Tunnicliffe DJ. Immunosuppressive treatment for primary membranous nephropathy in adults with nephrotic syndrome. Cochrane Database Syst Rev. 2021 Nov 15;11(11):CD004293. doi: 10.1002/14651858.CD004293.pub4. PMID 34778952